CLINICAL TRIAL: NCT00570375
Title: Phase II of Erlotinib an Epidermal Growth Factor Receptor Inhibitor in the Treatment of Myelodysplastic Syndrome
Brief Title: The Role of Erlotinib an Epidermal Growth Factor Receptor (EGFR) Inhibitor in the Treatment of Myelodysplastic Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution
Sponsor: University of Cincinnati (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07092512
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2009-04

CONDITIONS: Myelodysplastic Syndrome
Keywords: Blood disease, bone marrow
MeSH Terms: conditions — Myelodysplastic Syndromes; Hematologic Diseases | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): All patients will receive 150 mg of Erlotinib
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — 150 mg, PO, QD beginning day 1 week 1. Patients will receive treatment for 16 weeks as long as there is no evidence of disease progression. In no response is noted after 16 weeks of treatment, patients will be taken off the study. Patients achieving response (HI, CR, or PR) will continue on treatment until evidence of disease progression or relapse.
  Other Names: Tarceva®

SUMMARY:
The purpose of this research study is to find out what effects, good and/or bad, Erlotinib has on Myelodysplastic syndrome. Myelodysplastic syndrome is a group of blood diseases where the bone marrow (spongy space in long bones which is the factory for blood cell production) does not make enough blood cells and therefore there is a lack of healthy blood cells in the body. This can result in anemia, risk for infection and/or bleeding..

DETAILED DESCRIPTION:
MDS is a neoplastic clonal stem disorder characterized by bone marrow failure with cytopenia, dyslastic morphological features and tendency to progress to acute myeloid leukemia. It is estimated that MDS is the most common hematological malignancy in the USA. Several treatment options are available for MDS ranging from supportive care, growth factor use, chemotherapy, stem cell transplantation, and newer novel agents such as thalidomide, lenalidomide, and hypomethylating agents. Each of the different available treatments for MDS work in certain subset and relatively small percentage of patients, keeping the door open for novel therapeutic strategies to be explored. The NIH has published requests for applications on myeloproliferative and myelopdysplastic syndrome emphasizing the need for more research in this area.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an established diagnosis of myelodysplastic syndrome (MDS) and have either symptomatic anemia (defined as hemoglobin less than 10.0 g/dl) or transfusion dependent anemia (defined as 4 units of blood in the last 60 days).
* Patients treated previously with 5-azacytidine, decitabine, thalidomide, revlimid, amifostine, hydroxyurea, Histone deacytlase inhibitors and arsenic trioxide are allowed. Prior treatment with cytokines (i.e., interferon, interleukin), colony stimulating factors, or hydroxyurea is also permitted. Patients should be 28 days off prior treatment.
* Patients with chronic myelomonocytic leukemia (CMML) are eligible.
* Patients must have a performance status of 0 - 2 by Zubrod performance status criteria.
* Pretreatment pathology materials must be available for morphologic review. Collection of blood and marrow specimens for pathology review must be completed within 28 days prior to registration
* All patients must be informed of the investigational nature of this study and must sign and give written consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Patients must not have undergone bone marrow or stem cell transplant.
* Patients must not have received prior remission induction chemotherapy as treatment for MDS.
* Patients must not have secondary or therapy related MDS
* Patients who are known HIV positive are not eligible for this study.
* Patients must not be pregnant or nursing because of the potential risks of the drugs used in this study. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for at least 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
First 20 patients will be evaluated for overall response rate (CR, PR or HI). | Estimated to be about 1 year.

SECONDARY OUTCOMES:
If the first analysis of 20 patients warrant further enrollment, an additional 15 eligible patients will be registered. If 8 or more of the 35 patients achieve CR, PR or HI, then Phase III study will be warranted. | Estimated to be about 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Carl W Siegrist, M.D., Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- See also: University of Cincinnati Cancer Center — http://www.uccancercenter.uc.edu/